CLINICAL TRIAL: NCT00331916
Title: AL-15469A for the Treatment of Bacterial Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-04-38
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2009-09-29 (Estimated); Status verified 2009-09

CONDITIONS: Bacterial Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Bacterial | interventions — Quinolones

INTERVENTIONS:
Drug: quinolone

SUMMARY:
The purpose of the study is to determine whether AL-15469A is safe and effective in the treatment of bacterial conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Signs & Symptoms of conjunctivitis

Exclusion Criteria:

* Under 1 mo. age

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2005-11; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Clinical cure and microbiological success

SECONDARY OUTCOMES:
Individual signs and symptoms of bacterial conjunctivitis at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Stella Robertson, Ph.D., Study Director — Study Director
Locations (1):
- US, Fort Worth, Texas, United States